CLINICAL TRIAL: NCT03248960
Title: A Prospective Multi-Centre Study of the Ellume.Lab Flu A+B Test and iTreat Flu A+B Flu Test Performance Versus Viral Culture and Reverse Transcriptase Polymerase Chain Reaction.
Brief Title: Ellume.Lab Flu A+B Test and iTreat Flu A+B Flu Test Performance Versus Viral Culture and Reverse Transcriptase Polymerase Chain Reaction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ellume Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: iE-FLU-AUS-1701
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- iTreat Flu A+B Test and ellume.lab Flu A+B Test (Experimental): Upper respiratory tract samples from participants will be tested with:
  iTreat Flu A+B Test; ellume.lab Flu A+B Test; Reverse Transcriptase Polymerase Chain Reaction (RT-PCR); and viral culture.
  Interventions: Diagnostic Test: iTreat Flu A+B Test; Diagnostic Test: ellume.lab Flu A+B Test; Diagnostic Test: Reverse Transcriptase Polymerase Chain Reaction (RT-PCR); Diagnostic Test: Viral culture

INTERVENTIONS:
Diagnostic Test: iTreat Flu A+B Test — The iTreat Flu A+B Test is a rapid in vitro diagnostic test for the detection of influenza A or influenza B in nasal swab samples. The iTreat Flu A+B Test is designed to be simple to use and generates a result within 15 minutes.
Diagnostic Test: ellume.lab Flu A+B Test — The ellume.lab Flu A+B Test is an in vitro diagnostic test intended to be used at point-of-care for the detection of influenza A or influenza B in nasal swab samples. The ellume.lab Flu A+B Test generates a result within 10 minutes.
Diagnostic Test: Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) — Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) is a molecular diagnostic technique for the detection and identification of influenza viruses, both for clinical samples and isolates. The reverse transcriptase polymerase chain reaction (RT-PCR) allows template viral RNA to be reverse transcribed producing complementary DNA (cDNA) which can then be amplified and detected.
Diagnostic Test: Viral culture — Nasopharyngeal samples will be inoculated into appropriate culture media for influenza viral culture. In this test, the virus is actually grown and further identified in the laboratory as influenza A or B.

SUMMARY:
The primary purpose of this study is to validate the sensitivity and specificity of the iTreat Flu A+B Test and the ellume.lab Flu A+B Test in detecting influenza A and influenza B as compared to viral culture.

The secondary aims are to:

Validate the sensitivity and specificity of the iTreat Flu A+B Test and the ellume.lab Flu A+B Test in detecting influenza A and influenza B as compared to Reverse Transcriptase Polymerase Chain Reaction (RT-PCR).

Evaluate the correct interpretation of the iTreat Flu A+B Test by subjects with influenza-like symptoms.

Evaluate the subjects' satisfaction with the convenience, comfort and ease of use of the iTreat Flu A+B Test.

Evaluate the operators' satisfaction with the ease of use of the ellume.lab Flu A+B Test.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged ≥ 18 years: iTreat Flu A+B Test and ellume.lab Flu A+B Test OR aged ≥ 1 and <18 years: ellume.lab Flu A+B Test only; and
* Fever ≥ 37.8°C (100°F) at presentation or history or parent/guardian-reported history of fever ≥ 37.8°C (100°F) or feeling feverish within 24 hours of presentation; and
* Rhonorrhea or blocked nose; and
* Participant (or parent/legal guardian) capable and willing to give informed consent/assent; and
* Participant (or parent/legal guardian) able to read and write in English.

Exclusion Criteria:

* Participants aged <1 year.
* Participants who have undergone treatment with Tamiflu (oseltamivir), Relenza (zanamivir) or Symmetral (amantadine) within the previous 7 days.
* Participants who have been vaccinated by means of an influenza nasal spray/mist vaccine within the previous 7 days.
* Participants who have had a nose bleed within the past 30 days.
* Participants who have had recent craniofacial injury or surgery, including surgery to correct deviation of the nasal septum, within the previous 6 months.
* Participants currently enrolled in another clinical trial or have used any investigational device within 30 days preceding informed consent.
* Participants 18 years of age or older unable to understand English and consent to participation.
* Parent/legal guardian of Paticipants <18 years of age unable to understand English and consent to participation of child.
* Participants who have had prior exposure to iTreat Flu A+B Test.
* participants who have been previously enrolled in the iE-FLU-AUS-1701 study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2017-12-23 (Actual)

PRIMARY OUTCOMES:
Of participants positive for influenza A by viral culture, the percentage who are positive for influenza A by iTreat Flu A+B Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants positive for influenza A by viral culture, the percentage who are positive for influenza A by ellume.lab Flu A+B Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza A by viral culture, the percentage who are negative for influenza A by iTreat Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza A by viral culture, the percentage who are negative for influenza A by ellume.lab Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants positive for influenza B by viral culture, the percentage who are positive for influenza B by iTreat Flu A+B Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants positive for influenza B by viral culture, the percentage who are positive for influenza B by ellume.lab Flu A+B Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza B by viral culture, the percentage who are negative for influenza B by iTreat Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza B by viral culture, the percentage who are negative for influenza B by ellume.lab Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.

SECONDARY OUTCOMES:
Of participants positive for influenza A by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are positive for influenza A by iTreat Flu A+B Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants positive for influenza A by RT-PCR, the percentage who are positive for influenza A by ellume.lab Flu A+B Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza A by RT-PCR, the percentage who are negative for influenza A by iTreat Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza A by RT-PCR, the percentage who are negative for influenza A by ellume.lab Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants positive for influenza B by RT-PCR, the percentage who are positive for influenza B by iTreat Flu A+B Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants positive for influenza B by RT-PCR, the percentage who are positive for influenza B by ellume.lab Flu A+B Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza B by RT-PCR, the percentage who are negative for influenza B by iTreat Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza B by RT-PCR, the percentage who are negative for influenza B by ellume.lab Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Percent of participants who correctly interpret result of iTreat Flu A+B Test. | 1 day
  Agreement between trained staff and participants. Report as a percentage of participants with 95% confidence limits
Scores from questionnaire to assess ease of use, comfort and convenience of iTreat Flu A+B Test. | 1 day
  The ease of use questionnaire will provide total number of responses to each question and the percentage of participants selecting each response (on a 5 point Likert scale).
Scores from questionnaire to assess ease of use and convenience of ellume.lab Flu A+B Test. | 1 day
  The ease of use questionnaire will provide total number of responses to each question and the percentage of participants selecting each response (on a 5 point Likert scale).

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (8):
  - Ochre Health Medical Centre Casey, Casey, Australian Capital Territory
  - Paratus Clinical Blacktown Trial Clinic, Blacktown, New South Wales
  - Paratus Clinical Kanwal Trial Clinic, Kanwal, New South Wales
  - Coastal Family Health, Buddina, Queensland
  - Morayfield Family Doctors, Morayfield, Queensland
  - USC Health Clinics, Sippy Downs, Queensland
  - Griffith University Clinical Trial Unit, Southport, Queensland
  - Emeritus Research, Malvern East, Victoria